CLINICAL TRIAL: NCT00276185
Title: Effect of Botulinum Toxin Injections on Motor and Functional Ability of Upper Limb in Adults at Earlier Phases of Spastic Hemiplegia After Stroke
Brief Title: HEMITOX : Effect of Botulinum Toxin Injections on Motor and Functional Ability of Upper Limb in Adults at Earlier Phases of Spastic Hemiplegia After Stroke
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: J. Rebeyrol Hospital in Limoges (Unknown); Rennes University Hospital (Other); Center of Physical Medicine and Rehabilitation (Notre Dame de Lourdes Center in Rennes) (Unknown); Saint Jacques Hospital in Nantes (Unknown); Centre Hospitalier Universitaire de Saint Etienne (Other); Centre Régional de Département de médecine physique et réadaptation CHU-C3RF in Angers (Unknown); Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Pr Franck DURIF, CHU Clermont-Ferrand
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CHU63-0003
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Hemiplegia
Keywords: spasticity ;; Botulinum toxin ;; Upper limb ;; motor function.; spastic hemiplegia after stoke
MeSH Terms: conditions — Hemiplegia; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Time delay treatment of botulinum toxin

SUMMARY:
Botulinum toxin produced beneficial effects in spasticity in the hemiplegic upper limb. This study will test if botulinum toxin injections at earlier phases (<or = 3 months) in spasticity improve functional and motor tests compared with late injections (>or = 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 18
* Spastic hemiplegia after ischemic stroke (carotid occlusion) within the past 3 months.
* Antispasticity medication stabilized for the last 30 days
* Severe cognitive impairment such that patient is unable to provide scale assessment.
* Significant spasticity impeding improvement by re-education for 2 months or less
* Lack of muscular retraction defined by a minimal range of articular motion as :

  * finger : complete extension and rolling up
  * wrist : extension 40°/flexion : 45°
  * elbow : extension - 10°/flexion : 120°
  * shoulder : Enjalbert score 2 or more
* Antagonist muscles (to spasticity) activity score 1 or more
* Social Security benefits

Exclusion Criteria:

* Ischemic stroke thought to be due to basilar or vertebral vessel occlusion
* Known motor neuron or neuromuscular junction disease, disorders in which pain limits the ability to inject muscles (algodystrophy)
* Absence of mobility in proximal part of upper limb that does not predict a functional gain
* Minor stroke with non-disabling deficit or rapidly improving motor symptoms
* other serious illness, e.g. severe hepatic, cardiac, or renal failure ; acute myocardial infarction ; or a complex disease that may confound treatment assessment
* Treatment of spasticity by previous administration of botulinum toxin, if known
* Known allergy to botulinum toxin
* Currently participating in other research studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2005-12; Primary Completion 2009-01 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Deficiency, incapacity, handicap : Frenchay Arm test(post stroke arm function); Enjalbert test;
Box and blocks test
Enjalbert test
Modified Ashworth scale (upper limb)
Functional Independence Measure
Fugl-Meyer upper limb test
Clinical Global Impression (CGI)
36-Item Short Form (SF-36) quality of life

SECONDARY OUTCOMES:
Range of pain
Individual functional kinesitherapy

CONTACTS AND LOCATIONS:
Overall Officials: Franck Durif, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Result] Wissel J, Muller J, Dressnandt J, Heinen F, Naumann M, Topka H, Poewe W. Management of spasticity associated pain with botulinum toxin A. J Pain Symptom Manage. 2000 Jul;20(1):44-9. doi: 10.1016/s0885-3924(00)00146-9. PMID 10946168